CLINICAL TRIAL: NCT05410184
Title: The Effect of Virtual Reality Glasses and Application of Mural Curtain on Satisfaction, Tolerance, Comfort and Embarrassment During Colonoscopy
Brief Title: Effects of VR and Mural Curtain During Colonoscopy
Acronym: VR_COLON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Hasan Genç, Asistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: vr/curtain colon
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Misadventure During Endoscopic Examination
Keywords: virtual reality; tolerance; embarrassment; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: experimental model using randomized pretest and posttest with control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (Experimental): Except for the preparation of the patient for the procedure, since the colonoscopy procedure takes approximately 30 minutes, 30-minute 360-degree VR video scenes will be watched using the phone and VR head device.
  Interventions: Device: Virtual Reality Glasses group
- Mural Curtain (Experimental): the mural curtain group; they will be asked to focusing the mural curtain with a nature view during the colonoscopy procedure.
  Interventions: Other: mural curtain group
- control group (No Intervention): Patients of the control group, will not receive any intervention except for applied routine hospital colonoscopy procedures.

INTERVENTIONS:
Device: Virtual Reality Glasses group — Except for the preparation of the patient for the procedure, since the colonoscopy procedure takes approximately 30 minutes, 30-minute 360-degree VR video scenes will be watched using the phone and VR head device
  Arms: Virtual Reality Glasses
Other: mural curtain group — the mural curtain group; they will be asked to focusing the mural curtain with a nature view during the colonoscopy procedure.
  Arms: Mural Curtain

SUMMARY:
Background: Today, colonoscopy is widely used in many diseases, especially in the screening and diagnosis of colorectal cancers. Colonoscopy is considered a procedure that disturbs the patient's comfort because it is a very invasive and painful procedure. Along with physical discomfort during the procedure, it triggers emotional disturbances such as embarrassment, fear, and anxiety in the patient.

Purpose: To examine the effects of virtual reality glasses and video surveillance and picture screen application applied during colonoscopy on patients' satisfaction, tolerance, comfort and sense of shame.

Method: The population of the study consists of all patients who applied to Suleyman Demirel University Research and Practice Hospital, Department of General Surgery, Endoscopy Unit and were scheduled for colonoscopy. The sample will be represented by 180 patients whose colonoscopy procedure is planned between the specified dates and who meet the criteria for inclusion in the sample. In calculating the sample of the study, power analysis was performed and it was found the effect size of 0.40, 95% power and 0.01% margin of error for this study, that a total of 180 individuals for the three groups and at 60 individuals for each group. As a result, the sample of the research will consist of 180 people, 60 of whom are in the video with VR glasses, 60 people are in the mural curtain group and 60 people are in the control group. The study group of 180 people to participate in the study will be divided into three equal groups in accordance with the random numbers table obtained the computer-based Research Randomizer program. Data will be collected in the endoscopy unit on weekdays when the procedure is performed. The person who will collect the data is the endoscopy nurse working in the unit, one of the researchers. Colonoscopy procedure will be performed by the physician working in the unit, who is also one of the researchers. Before the colonoscopy procedure, the patients included in the study will be randomly divided into three groups: video group with VR, mural curtain group and control group. All participants in the study will first fill out a patient identification form containing patient demographic information. .

ELIGIBILITY:
Inclusion Criteria:

* 18 aged and over
* Written and verbal consent to participate in the study,
* Being conscious (person, place and time orientation),
* Undergoing colonoscopy for the first time

Exclusion Criteria:

* Having vision, hearing and communication problems
* Having any psychiatric and cognitive/mental mental health problems, disease (dementia, etc.),
* Diagnosed with visual, auditory and / or balance disorders,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-27 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | the fundamental characteristics of the patients will be filled in 15 minutes before the colonoscopy procedure
  This form, which was created by the researcher; Patients' age, gender, education level, marital status, employment status, income level, chronic disease status, previous surgery, complaints about coming to the hospital, having knowledge about colonoscopy, whether they would prefer the current method if they need to have colonoscopy again, It consists of a total of 14 questions questioning the use of additional sedation and painkillers during the procedure
Visual Analogue Scale (VAS) | Change from Baseline Visual Analogue Scale in 1 hour
  This scale developed by Price (1983) will be used in the research to determine the level of tolerance, comfort and satisfaction. It is a scale in which the distance between the two ends with a minimum value of 0 on one end and a maximum value of 10 on the other end is measured with a 10 cm ruler. In this context; The patient is explained that there are two endpoints and that he is free to mark any place between them that fits the severity of his pain. The distance between the beginning of "no comfort, tolerance and satisfaction" and this point marked by the patient is measured and recorded in centimeters. It has been shown that the VAS is a valid tool for the measurement of psychological and health variables such as pain and satisfaction, which is widely used in clinical studies (12).
The Colonoscopy Shame Scale | Change from Baseline The Colonoscopy Shame Scale in 1 hour
  this scale was developed in the United States in 2012 by Kimberly A. Mitchell and colleagues for the use of healthcare professionals. The scale consists of 15 questions examining the reasons why patients are ashamed of colonoscopy. For the statements in the scale, the participants mark the most appropriate answer for their own thoughts on a scale between 1 and 4 (strongly disagree=1, disagree=2, agree=3, totally agree=4). The lowest score that can be obtained from the total scale is 15, the highest score is 60. Higher scores indicate more embarrassment. The Cronbach's alpha coefficient of the original scale was 0.96. The validity and reliability study in Turkey was conducted by Koroglu in 2014 and the Cronbach's alpha coefficient of the scale was found to be 0.94 (11, 13).

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
all IPD that underlie results in a publication

REFERENCES:
- [Background] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Background] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- [Background] Bronner K, Mesters I, Weiss-Meilik A, Geva R, Rozner G, Strul H, Inbar M, Halpern Z, Kariv R. Determinants of adherence to screening by colonoscopy in individuals with a family history of colorectal cancer. Patient Educ Couns. 2013 Nov;93(2):272-81. doi: 10.1016/j.pec.2013.06.029. Epub 2013 Aug 2. PMID 23916675
- [Background] Umezawa S, Higurashi T, Uchiyama S, Sakai E, Ohkubo H, Endo H, Nonaka T, Nakajima A. Visual distraction alone for the improvement of colonoscopy-related pain and satisfaction. World J Gastroenterol. 2015 Apr 21;21(15):4707-14. doi: 10.3748/wjg.v21.i15.4707. PMID 25914482
- [Background] Veldhuijzen G, Klaassen NJM, Van Wezel RJA, Drenth JPH, Van Esch AA. Virtual reality distraction for patients to relieve pain and discomfort during colonoscopy. Endosc Int Open. 2020 Jul;8(7):E959-E966. doi: 10.1055/a-1178-9289. Epub 2020 Jun 30. PMID 32626819
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899